CLINICAL TRIAL: NCT05401877
Title: Factors Affecting Rehabilitation Time for Postoperative Complications Among Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE21096B
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: rehabilitation; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- short term rehabilitation: breast cancer survivors that recieved post-OP rehabilitation for equal or less than 300 minutes totally.
  Interventions: Procedure: therapies for breast cancer
- long term rehabilitation: breast cancer survivors that recieved post-OP rehabilitation for more than 300 minutes totally.
  Interventions: Procedure: therapies for breast cancer

INTERVENTIONS:
Procedure: therapies for breast cancer — the type of tumor removal surgery, combined therapy

SUMMARY:
Breast cancer patients who had undergone surgery, chemotherapy and radiotherapy suffered from complications, including shoulder stiffness, lymphedema and scar contracture. These symptoms impaired one's ADL function. Rehabilitation may relieved symptoms. However, it is difficult to estimate how long one should receive rehabilitation. The study is trying to establish a machine-learning based model in order to predict the period of rehabilitation.

DETAILED DESCRIPTION:
Breast cancer survivors suffered from complications after surgery, chemotherapy and radiotherapy. These complications include shoulder stiffness, upper limb lymphedema and scar contracture, which altogether impaired one's ADL function. Rehabilitation had been approved to relieved these symptoms effectively. However, many factor may interfere the patient's participation of rehabilitation, making it difficult to estimate how long one should receive rehabilitation. In Taiwan, National Health Insurance provides affordable, accessible and unlimited health care and medical service for all citizens, eliminating many social-economic barriers. Thus we are trying to establish a machine-learning based model in order to predict the period of rehabilitation.

Our study is a retrospective case-control study. The objectives are breast cancer survivors who attended post-surgery rehabilitation at least once for complications. The following data are collected from e-HIS system:

1. Patient characteristic: age, unilateral or bilateral cancer.
2. Surgery type: total, partial or simple mastectomy.
3. Lymphatic surgery: ALND and SLNB
4. Other surgical procedure: breast reconstruction, flap surgery.
5. Combined therapy: chemotherapy, radiotherapy or hormone therapy.
6. Complications: shoulder stiffness, lymphedema, scar contracture (ex., Axillary web syndrome), neurological deficit.
7. The first between operation and first time of rehabilitation.

The primary outcome is the total rehabilitation time, which will be divided as short term (less than 360 min) and long time (more than 360 min).

The data will be processed using WEKA and machine learning algorithms, including Logistic regression, supportive vector machine, K-nearest neighbors, decision tree and random forest.

ELIGIBILITY:
Inclusion Criteria:

* patients who received operation for breast cancer
* attended rehabilitation at least once for breast cancer related complications

Exclusion Criteria:

* patients who received rehabilitation for other reasons rather than surgical complications
* patients who are transfered to other hospital for rehabilitation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients that are registered at the case management system of Taichung Vetetans General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
the rehabilitation time | since the first session of rehabilitation until one year after the last session
  total post-operation rehabilitation time (minute)

CONTACTS AND LOCATIONS:
Overall Officials: Yuchun Lee, MD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No